CLINICAL TRIAL: NCT06510582
Title: Chronic Subdural Hematoma Treatment With Avastin® (Bevacizumab) Intra-Arterial Injection: A Non-Randomized, Open-Label Phase 1/2 Clinical Trial
Brief Title: Chronic Subdural Hematoma Treatment With Intra-Arterial Bevacizumab Injection
Acronym: CHAI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: Society of Vascular and Interventional Neurology (Unknown)
Responsible Party: Principal Investigator, Jane Khalife, MD, Assistant Professor of Neurology, The Cooper Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-154
Record Dates: First submitted 2024-06-28; First posted 2024-07-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Chronic intracranial subdural hematoma; Vascular endothelial growth factor; Bevacizumab; Middle meningeal artery embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Unilateral cSDH/ 2mg/kg Arm (Experimental): During phase 1, single 2mg/kg dose of bevacizumab to treat unilateral cSDH
  Interventions: Drug: Bevacizumab 2 mg/kg
- Phase 1 Bilateral cSDH/ 4mg/kg Arm (Experimental): During phase 1, two 2mg/kg doses (cumulatively 4mg/kg) of bevacizumab to treat bilateral cSDH
  Interventions: Drug: Bevacizumab 4 mg/kg
- Phase 2 Unilateral cSDH/ 2mg/kg Arm (Experimental): During phase 2, single 2mg/kg dose of bevacizumab to treat unilateral cSDH
  Interventions: Drug: Bevacizumab 2 mg/kg
- Phase 2 Bilateral cSDH/ 4mg/kg Arm (Experimental): During phase 2, two 2mg/kg doses (cumulatively 4mg/kg) of bevacizumab to treat bilateral cSDH
  Interventions: Drug: Bevacizumab 4 mg/kg

INTERVENTIONS:
Drug: Bevacizumab 2 mg/kg — Single 2mg/kg dose of bevacizumab to treat unilateral cSDH
  Arms: Phase 1 Unilateral cSDH/ 2mg/kg Arm; Phase 2 Unilateral cSDH/ 2mg/kg Arm
Drug: Bevacizumab 4 mg/kg — Two 2mg/kg doses (cumulatively 4mg/kg) of bevacizumab to treat bilateral cSDH
  Arms: Phase 1 Bilateral cSDH/ 4mg/kg Arm; Phase 2 Bilateral cSDH/ 4mg/kg Arm

SUMMARY:
The goal of this clinical trial is to test whether infusing bevacizumab into the middle meningeal arteries can be used to treat chronic subdural hematomas (cSDH).

The main questions it aims to answer are:

* Is bevacizumab infusion safe in cSDH patients?
* Is bevacizumab infusion effective in treating cSDH?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Radiographic evidence of chronic subdural hematoma, including

  1. Persistence of subdural blood more than 10 days after index traumatic injury or event
  2. Presence of mixed density blood
  3. Presence of subdural membranes
* Can obtain informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice contraception during participation in the study.
* Patients with concomitant intracranial pathology other than subdural hematoma (e.g., intracranial malignancy).
* Patients with known hypersensitivity to bevacizumab.
* Patients with radiographic evidence of mass effect.
* Patients have focal neurological deficits attributed to subdural hematoma.
* Patient had craniotomy or burr hole operative procedures performed in preceding two weeks prior to onset of subdural hematoma.
* Secondary causes apart from trauma for the chronic subdural hematoma, such as underlying vascular abnormality or tumor.
* Emergent surgical evacuation is required for the patient.
* Non-convexity chronic subdural hematoma, as the middle meningeal artery will not supply this area.
* Coagulation abnormalities, including platelet count <100,000 and/or international normalized ratio of <1.5 despite attempts for correction.
* Patients with known contraindications for angiography. Patients with contrast allergy will be premedicated with diphenhydramine and steroids.
* Patient has known active systemic infection or sepsis.
* Patient has contradiction to anesthetic agents used for conscious sedation/monitored anesthesia care (MAC).
* Patient has life expectancy of less than six months due to comorbid terminal conditions.
* Patient has a premorbid modified Rankin score (mRS) of 5 or greater.
* Concurrent participation in another research protocol for investigation of an experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events | Up to 3 months after study treatment
  Reported serious adverse events classified using MedDRA and CTCAE, in addition to treatment-related events and all other adverse events

SECONDARY OUTCOMES:
Rate of Hematoma Recurrence | 3 months after study treatment and 6 months after study treatment
  Rate of hematoma recurrence or progression requiring intervention and/or readmission
Rate of Complete Hematoma Resolution | 3 months after study treatment and 6 months after study treatment
  Rate of complete hematoma resolution compared to baseline on imaging
Rate of Partial Hematoma Resolution | 3 months after study treatment and 6 months after study treatment
  Rate of at least 50% or greater reduction in hematoma size from baseline on imaging
Change in Hematoma Size | 3 months after study treatment and 6 months after study treatment
  Change in hematoma size measured in millimeters on imaging
Change in Clinical Neurological Symptom Scale Scores: NIHSS | 3 months after study treatment and 6 months after study treatment
  Change in National Institutes of Health Stroke Scale (NIHSS) scores, scores range from 0 to 42, with higher scores indicating more severe neurological deficit
Change in Clinical Neurological Symptom Scale Scores: GCS | 3 months after study treatment and 6 months after study treatment
  Change in Glasgow Coma Scale (GCS) scores, ranging from 3 to 15 with lower score indicating more impaired consciousness
Change in Clinical Neurological Symptom Scale Scores: mRS | 3 months after study treatment and 6 months after study treatment
  Change in modified Rankin Scale (mRS) scores, ranges from 0-6 with higher score indicating worse functional outcome

OTHER OUTCOMES:
Number of Participants with Anatomical Variants | During the treatment procedure
  Middle meningeal arteries with dangerous anastomoses observed on imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jane Khalife, MD, Principal Investigator — The Cooper Health System; Ajith J Thomas, MD, Study Chair — The Cooper Health System; Manisha Koneru, MD, Study Chair — The Cooper Health System
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

REFERENCES:
- [Background] Khalife J, Tonetti DA, Shaikh H, Jovin T, Patel P, Thomas A. Intraarterial bevacizumab administration through the middle meningeal artery for chronic subdural hematoma. Stroke: Vascular and Interventional Neurology. 2023 Jul;3(4). doi:10.1161/svin.122.000722
- [Background] Khalife J, Koneru M, Tonetti DA, Shaikh HA, Jovin TG, Patel PD, et al. Intra-arterial selective bevacizumab administration in the middle meningeal artery for chronic subdural hematoma: An early experience in 12 Hemispheres. Stroke: Vascular and Interventional Neurology. 2024 Sept;4(5). doi:10.1161/svin.124.001409